CLINICAL TRIAL: NCT05927246
Title: Radiotherapy-associated Atrial Fibrillation: Onset Time and Frequency
Brief Title: Radiotherapy-Associated Atrial Fibrillation
Acronym: RADAF
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Cafer Zorkun, Head, Division of CardioOncology, Istanbul University
Other Study IDs: COEXIST-1
Record Dates: First submitted 2023-06-23; First posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Atrial Fibrillation New Onset
Keywords: Atrial fibrillation; breast cancer; lung cancer; thoracic malignancies; cardiotoxicity
MeSH Terms: conditions — Atrial Fibrillation; Breast Neoplasms; Lung Neoplasms; Cardiotoxicity | interventions — Electrocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Thoracic Malignancies: All patients undergoing RT for Thoracic Malignancies
  Interventions: Diagnostic Test: ECG
- Patients with Breast Cancer: All patients undergoing RT for Breast Cancer
  Interventions: Diagnostic Test: ECG

INTERVENTIONS:
Diagnostic Test: ECG — 12 lead ecg for each participant

SUMMARY:
Radiotherapy associated Atrial Fibrillation (RADAF) is an observational study to evaluate onset time and frequency of atrial fibrillation in patients with thoracic malignancies and breast cancer.

Each patient will have 12 lead ECG prior, and daily during radiotherapy.

DETAILED DESCRIPTION:
Collected data will be truly anonymised and individuals will no longer identifiable, and than evaluated for occurrence of atrial fibrillation.

Inclusing Criteria:

1. Patients with radiotherapy for thoracic malignancy or breast cancer
2. Between 18-99 years-old

Exclusion Criteria:

1. Patients with history of radiotherapy
2. Patients with history of atrial fibrillation
3. Patients with pacemaker implantation

ELIGIBILITY:
Inclusion Criteria:

* Patients with radiotherapy for thoracic malignancy or breast cancer
* Between 18-99 years-old

Exclusion Criteria:

* Patients with history of radiotherapy
* Patients with history of atrial fibrillation
* Patients with pacemaker implantation

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with breast and thoracic cancers will be evaluated for incidence and onset time of AFib.
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Occurrence of atrial fibrillation | 1 day During radiotherapy
  Occurrence of atrial fibrillation
Onset time of atrial fibrillation | 1 day During radiotherapy
  Onset time of atrial fibrillation

CONTACTS AND LOCATIONS:
Overall Officials: Cafer Zorkun, MD PhD, Principal Investigator — Faculty member
Locations (1):
- Istanbul Faculty of Medicine, Fatih, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No